CLINICAL TRIAL: NCT04086303
Title: Is There Any Difference in Anthropometric and Physical Fitness Parameters in Handball Players?
Brief Title: Anthropometric and Physical Fitness Differences Among Turkish Adolescents and Adults Handball Players
Acronym: Handball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guven Health Group (Other)
Responsible Party: Principal Investigator, GUL BALTACI, PROFESSOR, PT.PH.D., Guven Health Group
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 520
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Athletic Performance; Physical Fitness; Handball Players; Cross-sectional Studies
MeSH Terms: interventions — 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid

STUDY DESIGN:
Intervention Model Description: young handball players ≥10 years sport age adult handball players ≤10 years sport age
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- young handball players (Experimental): The first group was named young players (n = 19; age = 18.05 ± 2.58 years, body mass index = 22.0 ± 2.21 kg, sport participation ≤ 10 years)
  Interventions: Other: LSST test
- adult handball players (Active Comparator): The second group was named old players (n =23; age = 28,91 ± 3.39 years, body mass index = 22.20 ± 2.75 kg, sport participation ≥ 11 years).
  Interventions: Other: LSST test

INTERVENTIONS:
Other: LSST test — LSST test: Scapular mobility testing Upper Extremity test: Upper extremity agility and endurance testing Y Balance test: Balance and Coordination testing Sit and Reach Test: Assessment of flexibility
  Other Names: upper extremity test; Y Balance test; Sit and reach test

SUMMARY:
The purpose of this study was to examine the variation in physical and physiological characteristics according to sports age in adolescent and adult male team handball (TH) players. Adolescent (N.=19, aged 18.1±1.4 yr) and adult (N.=23, 28.6±5.7 yr) players were examined for anthropometric characteristics, somatotype and body composition, and performed the physical working capacity test, a force-velocity test, the lateral scapular slide test (LSST), shark skill test, Davies test, squat jump (SJ), countermovement vertical jump without (CMJ).

DETAILED DESCRIPTION:
The stability of the scapula in relation to the entire moving upper extremity is the key in the throwing sequence. The importance of scapular positioning in handball players has been well documented in the literature, but no one has compared scapular positioning between handball players and sedentary people. Study participants completed a rating scale for pain and a questionnaire about demographic and shoulder problems. One assessor performed the lateral scapular slide test and additional flexibility measurements around the shoulder girdle. Flexibility (external rotation, internal rotation) and scapular position (1, 2, 3) were compared among groups (young players, old players, sedentary people) and between sides (dominant, nondominant).

Participants: Forty-five aged between 16 and 35 yrs were recruited in the study. The exclusion criteria included those (a) with soft tissue or bone problems affecting lower and upper extremity, (b) who had acute inflammation affecting upper and lower extremity region, (c) had scoliosis, (d) who had undergone any orthopedic surgery, (e) who had defined any pain or painful area at lower extremities and (f) who were obese (BMI>30 kg/m2).

Assessments: The investigators plan to perform the physical working capacity test, a force-velocity test, the lateral scapular slide test (LSST), shark skill test, Davies test, squat jump (SJ), countermovement vertical jump without (CMJ).

The power analysis indicated that 32 participants for total were needed with 80 % power and a 5 % type 1 error. The power analysis of our study showed a power of 80% with LSST as the primary outcome. The data were analyzed using statistical software (SPSS version 18, Inc., Chicago, IL, USA). All the statistical analyses were set a priori at an alpha level of p<0.05. The tests for homogeneity (Levene's test) and normality (Shapiro-Wilk) were used to determine the appropriate statistical methods. According to the test results, nonparametric Friedman test was used for comparisons between baseline, first taping and last taping. Wilcoxon test was used for possible differences which may occur between taping applications in order to identify the application that provided the difference. Parametric test assumptions were not possible due to small sample size and inhomogeneous parameters.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were the ability to actively perform pain-free abduction from 0° to 45° and from 0° to 90° in elbow extension and age greater than 15 years.
* to be volunteer for including the study
* to be ready mentally

Exclusion Criteria:

* Exclusion criteria were shoulder injury, shoulder surgery in the 2 years before the study, systemic pathologic condition, or intervention in the 3 months before the study, including corticosteroid or hydrodilatation injection or physiotherapy.
* Specifically, injury included shoulder pain in active abduction or external rotation for more than 3 months, a reason to suspect a complete rotator cuff tear (eg, substantial shoulder weakness), a positive drop-arm sign or previous fracture, or a high-riding humerus observed on plain radiographs.
* Systemic pathologic conditions included inflammatory joint disease, complex regional pain syndrome, and shoulder pain referred from vertebral structures that was diagnosed via spinal clearing tests.

Ages: 16 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — having only male handball players
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Testing for LSST | 30 minutes
  To maintain a consistent posture during the various test positions, participants were instructed to fix their eyes on an object in the examination area. For test position 1 of the LSST, participants were instructed to keep their upper extremities relaxed at their sides. The assessor obtained and confirmed the test position and then identified through palpation and marked the inferior aspect of the inferior angle of the scapula and the closest spinous process in the same horizontal plane.
Upper extremity Test (Davies test) | 30 minutes
  Place 2 pieces of tape on the floor 90 cm apart, in a push up position with one hand on each tape. Have the client touch the other hand and alternate for 15 seconds. Repeat 3 times.
Y Balance Test | 15 minutes
  The athlete should be wearing lightweight clothing and remove their footwear. After doing so, they are the required to stand on centre platform, behind the red line, and await further instruction.
Sit and Reach Test | 10 minutes
  The test evaluates flexibility. Subjects are seated with their legs joined and outstretched. The soles of their feet are supported in a standardised wood box (Well Box). Through inflection of their trunks, the subjects reach (with their ring fingers, arms joined and hands superposed) as far as they can toward/upon the box; they perform this reaching movement 2 times, and the maximal distance is recorded. The accuracy of this measurement in the present study is to within 0.1 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Sardan Cetinkaya, MD, Study Director — Guven Health Group
Locations (1):
- Guven Health Group, Ankara, Turkey (Türkiye)